CLINICAL TRIAL: NCT02805478
Title: Fat-Associated Cardiovascular Organ Dysfunction
Acronym: FATCOR
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 189.08
Record Dates: First submitted 2016-06-12; First posted 2016-06-20 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-04

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The FATCOR Research biobank has been approved by Health authorities and includes samples from serum, whole blood, urine
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: There is no intervention — This is a prospective observational cohort study without any intervention

SUMMARY:
This is an observational study of cardiovascular risk factors and arterial or cardiac function in subjects with overweight or obesity. Subjects must be between 30 and 65 years of age, have a body mass index >27.0 kg/m2 and free from known heart disease and digestive or psychiatric disorders. Study aims include identifying sex-differences in traditional cardiovascular risk factors and structural and functional abnormalities in arteries and the heart in subjects with overweight or obesity, and how this is influenced by physical fitness.

DETAILED DESCRIPTION:
FATCOR is an observational study of women and men with overweight or obesity. In particular prevalences of conventional cardiovascular risk factors and subclinical arterial or cardiac dysfunction are explored. The study aims at identifying sex differences in presence and clustering of cardiovascular risk factors and presence of subclinical cardiovascular organ damage. The influence of physical fitness on these factors will also be assessed. All participants undergo extensive cardiovascular risk factor assessment including oral glucose tolerance test and ambulatory blood pressure recording. Subclinical cardiovascular dysfunction is assessed by carotid and femoral vascular ultrasound, echocardiography and carotid-femoral pulse wave velocity using applanation tonometry. Physical fitness is assessed from peak oxygen uptake during maximal exercise testing on a treadmill.

ELIGIBILITY:
Inclusion Criteria:

* body mass index > 27.0 kg/m2

Exclusion Criteria:

* known heart disease
* digestive disorder
* psychiatric disorder
* unfamiliar with Norwegian language

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Norwegian women and men
Sampling Method: Non-Probability Sample
Enrollment: 618 (Actual)
Dates: Start 2009-09-05 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Abnormal left ventricular geometry | At study baseline
  Echocardiography
Dilated left atrium | At study baseline
  Echocardiography

SECONDARY OUTCOMES:
Relation of physical fitness to prevalence of cardiovascular risk factors | At study baseline
  Cardiopulmonary exercise
Relation of sex to prevalence of hypertension | At study baseline
  Ambulatory blood pressure recording
Relation of sex to abnormal left ventricular geometry | At study baseline
  Echocardiography
Relation of sex to arterial stiffness | At study baseline
  Applanation tonometry

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Vikenes, MD PhD, Study Director — Haukeland University Hospital, Department of Heart Disease
Locations (1):
- Haukeland University Hospital, Department of Heart Disease, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Halland H, Lonnebakken MT, Saeed S, Midtbo H, Cramariuc D, Gerdts E. Does fitness improve the cardiovascular risk profile in obese subjects? Nutr Metab Cardiovasc Dis. 2017 Jun;27(6):518-524. doi: 10.1016/j.numecd.2017.04.006. Epub 2017 Apr 26. PMID 28528703
- [Result] Halland H, Lonnebakken MT, Pristaj N, Saeed S, Midtbo H, Einarsen E, Gerdts E. Sex differences in subclinical cardiac disease in overweight and obesity (the FATCOR study). Nutr Metab Cardiovasc Dis. 2018 Oct;28(10):1054-1060. doi: 10.1016/j.numecd.2018.06.014. Epub 2018 Jun 21. PMID 30177273
- [Result] Halland H, Matre K, Einarsen E, Midtbo H, Saeed S, Pristaj N, Lonnebakken MT, Gerdts E. Effect of fitness on cardiac structure and function in overweight and obesity (the FATCOR study). Nutr Metab Cardiovasc Dis. 2019 Jul;29(7):710-717. doi: 10.1016/j.numecd.2019.03.012. Epub 2019 Apr 3. PMID 31138499
- [Derived] Midtbo H, Ulvik A, Cramariuc D, Meyer K, Ueland PM, Halland H, Gerdts E. Influence of cardiorespiratory fitness on obesity-associated inflammation in women and men: The FATCOR study. Nutr Metab Cardiovasc Dis. 2024 Aug;34(8):1942-1949. doi: 10.1016/j.numecd.2024.04.002. Epub 2024 Apr 12. PMID 38749786
- [Derived] Pristaj N, Saeed S, Midtbo H, Halland H, Matre K, Gerdts E. Covariables of Myocardial Function in Women and Men with Increased Body Mass Index. High Blood Press Cardiovasc Prev. 2020 Dec;27(6):579-586. doi: 10.1007/s40292-020-00418-6. Epub 2020 Oct 24. PMID 33098553
- [Derived] Herfindal B, Gerdts E, Kringeland EA, Saeed S, Midtbo H, Halland H. Concomitant hypertension is associated with abnormal left ventricular geometry and lower systolic myocardial function in overweight participants: the FAT associated CardiOvasculaR dysfunction study. J Hypertens. 2020 Jun;38(6):1158-1164. doi: 10.1097/HJH.0000000000002397. PMID 32371806